CLINICAL TRIAL: NCT06383832
Title: Effect of Dapagliflozin on Body Weight in Overweight Women Consuming Different Proportions of Carbohydrate Diet.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Jia (Other)
Responsible Party: Sponsor-Investigator, Sun Jia, Chief Physician, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240310_GY
Record Dates: First submitted 2024-03-13; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Overweight; Carbohydrate; Sodium-glucose Transporter 2 Inhibitors
MeSH Terms: conditions — Overweight | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: This study included a total sample size of 36 subjects and underwent a 12 week intervention with dapagliflozin. Then, subgroup analysis was conducted. According to the 24-hour dietary review method on the 3rd day of each week during the introduction period, the low carbohydrate group accounted for 10-25% of the total energy intake due to carbohydrates, while the non low carbohydrate group accounted for 26% or more of the total energy intake due to carbohydrates.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dapagliflozin (Experimental): Dapagliflozin tablets oral 10mg/d qd. Treatment course:12 weeks. Then, subgroup analysis was conducted. According to the 24-hour dietary review on the 3rd day of each week during the introduction period, subjects with carbohydrate energy greater than or equal to 26% of their daily energy intake were included in the non low carbohydrate group (NCD group), while subjects with carbohydrate energy accounting for 10-25% of their daily energy intake were included in the low carbohydrate group (LCD group).
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin tablets oral 10mg/d qd, intervention for 12 weeks.

SUMMARY:
In recent years, the prevalence of overweight and obesity has increased dramatically worldwide, of which 34.3% and 16.4% of adults in China are overweight and obese, respectively, ranking first in the world's obese population. Dapagliflozin is a sodium-glucose transporter 2 Inhibitors that inhibits glucose reabsorption and promotes urinary glucose excretion by inhibiting renal proximal tubular sodium-glucose transporter 2 Inhibitors for the treatment of type 2 diabetes mellitus. The urinary glucose excretion induced by dapagliflozin can induce weight loss through energy loss or body water loss caused by osmotic diuresis. In addition, in patients with type 2 diabetes, dapagliflozin may also induce weight loss by reducing body fat as well as subcutaneous and visceral fat.In a randomized controlled trial, type 2 diabetes patients treated with sodium-glucose transporter 2 Inhibitors lost approximately 1-3 kg. Also, sodium-glucose transporter 2 Inhibitors have shown good weight loss in obese people without type 2 diabetes. In real-world studies, a minority of type 2 diabetes patients taking dapagliflozin experienced weight gain. The American Lipid Association defines a low carbohydrate diet as the calorie intake of carbohydrates accounting for 10-25% of the total daily energy intake. In a randomized controlled trial, a low-carbon diet showed a more significant decrease in body weight, fat mass index, whole body fat, and visceral fat after 8 weeks compared to the standard diet. So, this study intends to investigate whether the weight loss effect of dapagliflozin is affected by different dietary structures.

DETAILED DESCRIPTION:
Record the following indicators before and after intervention, including height, weight, BMI, blooAccording to previous literature, dapagliflozin has a weight loss effect on overweight/obese individuals. This study is a prospective, open label, single arm, exploratory clinical trial, expected to include 36 overweight women. The subjects enter a 4-week introduction period, during which they need to maintain their original dietary habits and record a 24-hour dietary review on the 3rd of each week. At the end of the introduction period, if the weight change of the subject is less than 3%, it is considered qualified. Then, qualified subjects will receive a 12 week intervention with dapagliflozin tablets (oral, 10mg, once a day). During the experiment, participants were required to maintain their original dietary habits unchanged. Participants are required to record their dietary habits for three days a week in order to determine their energy intake and carbohydrate energy ratio. d pressure, waist circumference, abdominal circumference, waist to hip ratio, morning urine routine, 24-hour urine glucose, fasting blood glucose, fasting insulin, blood lipids (TG/TC/LDL/HDL), body fat percentage, body fat mass, muscle mass, subcutaneous fat, visceral fat volume, and abdominal fat volume, and record any adverse reaction events that occurred during the study. Collect patient urine and serum samples for testing. Collect patient feces, freeze the samples in a -80 ℃ freezer, and send the feces to a biological company for testing of intestinal microbiota composition.

Conduct subgroup analysis, based on the 24-hour dietary review provided by the subjects on the 3rd day of the week during the introduction period, subjects with carbohydrate energy greater than or equal to 26% of their daily energy intake will be included in the non low carbohydrate group (NCD group), and subjects with carbohydrate energy accounting for 10-25% of their daily energy intake will be included in the low carbohydrate group (LCD group).

ELIGIBILITY:
Inclusion Criteria:

* Women.
* Age 18-45 years.
* 23.9kg/m2< BMI<28kg/m2.
* Less than 60 minutes of light activity per week.
* No contraindications to MRI.
* Voluntary participation and willingness to sign informed consent.

Exclusion Criteria:

* The weight change in the past three months is greater than 5%.
* Taking any medications or dietary supplements in the past 3 months that would affect weight/energy expenditure.
* Systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure≥ 90 mmHg.
* Including endocrine disorders such as diabetes and hyperthyroidism.
* Patients with the presence of acute/chronic infections, heart, liver, lung and kidney diseases.
* Alcoholism, smoking, strenuous exercise in the past 3 months.
* History of recurrent urinary tract infections.
* History of malignancy.
* Severe renal insufficiency, severe hepatic insufficiency.
* Patients who are pregnant, planning to become pregnant in the near future, or breastfeeding.
* Those with other conditions that prevent them from participating in the completion of the intervention follow-up.
* Participation in other clinical trials within the past 4 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Changes in Body mass index (BMI) i | At 12th week after the intervention.
  When measuring height, the subjects are required to take off their shoes, hats, and coats, keep their feet together in an upright position, keep their shoulders, head, and heels close to the ruler, and look straight ahead with the right-angle plate close to the top of the head. The measurement standard of height is accurate to 0.1cm. When measuring body weight, the subjects are required to take off their shoes, hats, and single clothes for measurement and the measurement standard of body weight is accurate to 0.1kg. Body mass index (BMI) is calculated by dividing body weight (kg) by the square of height (m2). All measurements will be performed by trained staff.

SECONDARY OUTCOMES:
Changes in fasting blood glucose. | At 12th week after the intervention.
  Fasting blood glucose will be uniformly implemented in the Laboratory.
Changes in waist circumference. | At 12th week after the intervention.
  When measuring the waist circumference, the subjects were required to wear thin underwear, and the researchers used a soft ruler to measure the midpoint of the line connecting the highest point of the iliac crest and the lower edge of the 12th rib around the abdomen in the horizontal direction, and the measurement of waist circumference was accurate to 0.1cm. All measurements are performed by trained staff.
Changes in insulin resistance index. | At 12th week after the intervention.
  The steady-state model assessment method will be used to calculate homeostasis model assessment of insulin resistance.
Changes in waist-to-hip ratio. | At 12th week after the intervention.
  When measuring the waist circumference, the subjects were required to wear thin underwear, and the researchers used a soft ruler to measure the midpoint of the line connecting the highest point of the iliac crest and the lower edge of the 12th rib around the abdomen in the horizontal direction, and the measurement of waist circumference was accurate to 0.1cm. When measuring the hip circumference, the subjects are required to wear thin underwear, and a soft ruler is required to measure the circumference of the most protruding part backwards around the buttocks to the nearest 0.1cm. The waist-to-hip ratio is calculated by dividing the waist circumference by the hip circumference. All measurements are performed by trained staff.
Changes in abdominal circumference. | At 12th week after the intervention.
  When measuring the abdominal circumference, the subjects were required to wear thin underwear and measured the circumference around the abdomen with a soft tape through the point of the iliac crest, measured to an accuracy of 0.1 cm.
Changes in Blood triglycerides | At 12th week after the intervention.
  will be tested by the Laboratory.
Changes in total cholesterol | At 12th week after the intervention.
  will be tested by the Laboratory.
Changes in low-density lipoprotein、high-density lipoprotein | At 12th week after the intervention.
  will be tested by the Laboratory.
Changes in body fat percentage. | At 12th week after the intervention.
  Body fat percentage will be tested using an body composition analyzer manufactured in Korea. Before the measurement, the subjects will be required to have an empty stomach and instructed to empty their urine and bowels. The subjects will be asked to use 75% alcohol gauze to wipe their hands and feet to make them fully contact the electrode surface of the analyzer after taking off their socks. Then researchers having training before will enter the patient's personal information on the body composition analyzer computer, and press the finish and start buttons next to get the body fat percentage measurement result.
Changes in subcutaneous fat volume. | At 12th week after the intervention.
  Specialized researchers used Dutch made Philips magnetic resonance imaging to scan the abdomen and upper part of the pelvis of the subjects. The scanning was performed using body coils, and after a period of adaptation, the subjects were scanned in a fixed ambient temperature in the scanning room. Based on the open-source image processing software from Harvard Medical School in the United States, semi-automatic image segmentation is performed on fat images to obtain subcutaneous fat volume, respectively; Based on open-source image processing software in the United States, the average value represents the fat fraction of the liver.
Changes in body fat volume. | At 12th week after the intervention.
  Body fat volume will be tested using an body composition analyzer manufactured in Korea. Before the measurement, the subjects will be required to have an empty stomach and instructed to empty their urine and bowels. The subjects will be asked to use 75% alcohol gauze to wipe their hands and feet to make them fully contact the electrode surface of the analyzer after taking off their socks. Then researchers having training before will enter the patient's personal information on the body composition analyzer computer, and press the finish and start buttons next to get the body fat volume measurement result.
Changes in the relative abundance of gut microbiota. | At 12th week after the intervention.
  At baseline and at the end of the trial, researchers will collect fecal samples from participants, all of which will be frozen and stored in a refrigerator. After the experiment, the fecal samples will be sent to Hangzhou Lianchuan Biotechnology Co., Ltd. to extract total fecal DNA. 16S rDNA sequencing technology will be used to detect the relative abundance of intestinal microorganisms.
Changes in urine. | At 12th week after the intervention.
  Morning urine routine、24h urine glucose will be uniformly implemented in the Laboratory.
Changes in β-hydroxybutyric acid. | At 12th week after the intervention.
  β-hydroxybutyric acid will be implemented in the Laboratory.
Changes in muscle mass. | At 12th week after the intervention.
  Muscle mass will be tested using an body composition analyzer manufactured in Korea. Before the measurement, the subjects will be required to have an empty stomach and instructed to empty their urine and bowels. The subjects will be asked to use 75% alcohol gauze to wipe their hands and feet to make them fully contact the electrode surface of the analyzer after taking off their socks. Then researchers having training before will enter the patient's personal information on the body composition analyzer computer, and press the finish and start buttons next to get the muscle mass measurement result.
Changes in fasting insulin. | At 12th week after the intervention.
  Fasting blood glucose、fasting insulin will be uniformly implemented in the Laboratory.
Changes in visceral fat volume. | At 12th week after the intervention.
  Specialized researchers used Dutch made Philips magnetic resonance imaging to scan the abdomen and upper part of the pelvis of the subjects. The scanning was performed using body coils, and after a period of adaptation, the subjects were scanned in a fixed ambient temperature in the scanning room. Based on the open-source image processing software from Harvard Medical School in the United States, semi-automatic image segmentation is performed on fat images to obtain visceral fat volume, respectively; Based on open-source image processing software in the United States, the average value represents the fat fraction of the liver.
Changes in hip circumference. | At 12th week after the intervention.
  When measuring the hip circumference, the subjects are required to wear thin underwear, and a soft ruler is required to measure the circumference of the most protruding part backwards around the buttocks to the nearest 0.1cm. The waist-to-hip ratio is calculated by dividing the waist circumference by the hip circumference. All measurements are performed by trained staff.
The incidence of adverse events. | At 12th week after the intervention.
  The investigator will ask participants in face-to-face visits or contacted with them by phone to record observed side effects and adverse events in time.

CONTACTS AND LOCATIONS:
Overall Officials: jia sun, MD,PhD, Study Chair — Zhujiang Hospital; jitong li, MD,PhD, Principal Investigator — Zhujiang Hospital
Locations (2):
- China (2):
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No